CLINICAL TRIAL: NCT03169881
Title: Darbepoetin Trial to Improve Red Cell Mass and Neuroprotection in Preterm Infants
Acronym: Darbe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0058
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Neurocognitive; Neuroprotective; Neonatal; Neurodevelopmental Impairment
MeSH Terms: interventions — Darbepoetin alfa; Saline Solution; Organization and Administration

STUDY DESIGN:
Intervention Model Description: Randomized, masked, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Primary providers and bedside caregivers will be blinded to randomization group. If the dose will be administered IV, the study drug will be administered slow IV push by the bedside nurse. If the dose will be administered subcutaneously, the study drug will be brought to the bedside in a closed container, and injections will be shielded behind screens and out of earshot from caregivers and parents. An adhesive bandage (or 2x2 gauze) will be placed over the true and sham injection sites and either taped or held in place until no evidence of the injection is visible. The parents, medical providers, data collection staff and neurodevelopmental follow up personnel will be masked to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darbepoetin (Experimental): Darbepoetin 10 micrograms/kg/once every week (IV or SC)
  Interventions: Drug: Darbepoetin
- Placebo (Placebo Comparator): Equal volume normal saline for IV administration, or sham dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin — Darbepoetin 10 micrograms/kg/once every week (IV or SC). Infants will be treated until 35 completed weeks gestation, discharge, or transfer to another hospital.
  Other Names: Darbe
  Arms: Darbepoetin
Drug: Placebo — normal saline for IV administration, or sham dosing. Infants will be treated until 35 completed weeks gestation, discharge, or transfer to another hospital.
  Other Names: normal saline for IV administration, or sham dosing
  Arms: Placebo

SUMMARY:
Study Hypothesis: Preterm infants administered weekly Darbe during the neonatal period will have improved neurocognitive outcome at 22-26 months compared to placebo

DETAILED DESCRIPTION:
Advances in neonatal care have led to significant improvements in the survival of the nearly 60,000 very low birth weight (VLBW) infants born each year in the U.S. Improving neurodevelopmental outcomes for these preterm infants continues to be a major goal for neonatal care providers. A subset of these infants sustain a grade 3 or 4 intraventricular hemorrhage (IVH) resulting in an increase in the incidence of developmental delay. Moreover, almost one third of preterm infants with normal head ultrasounds also develop cognitive delay. Although a variety of neuroprotective treatment strategies have been evaluated, no specific treatment has been identified to reduce or prevent brain injury in these most vulnerable preterm infants.

A potential neuroprotective therapy involves administering erythropoiesis stimulating agents (ESAs) such as erythropoietin (Epo) and Darbepoetin (Darbe, a longer acting ESA). In addition to stimulating erythropoiesis, ESAs have been shown to be protective in the developing brain in animal models, making it possibly beneficial for very premature infants who are at risk for intraventricular hemorrhage, hypoxic-ischemic injury, and developmental delay. The neuroprotective mechanisms of ESAs include increased neurogenesis, decreased neuronal susceptibility to glutamate toxicity, decreased neuronal apoptosis, decreased inflammation, decreased nitric oxide-mediated injury, increased antioxidant response, decreased axonal degeneration, and increased protective effects on glia. This is a randomized, masked, placebo controlled clinical study in which enrolled infants will receive weekly Darbe or placebo (sham) dosing.

Extended follow-up: Subjects will be seen for follow-up at 4-5 years (i.e., 4 years - 4 years 11 months) corrected age and 6-7 years (i.e., 6 years - 6 years 11 months) corrected age to characterize the functional, behavioral and neurological outcomes of the extremely low birth weight (ELBW) population at school age based on treatment with darbepoetin versus placebo in the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

* Inborn and outborn preterm infants
* 23 0/7-28 6/7 weeks gestational age
* ≤24 hours postnatal age

Exclusion Criteria:

* Hematocrit > 60%
* Infants with known congenital or chromosomal anomalies, including congenital heart disease and known brain anomalies
* Hemorrhagic or hemolytic disease
* EEG- confirmed seizures
* Congenital thrombotic disease
* Systolic blood pressures >100 mm Hg while not on pressor support
* Receiving Epo or Darbe clinically, or planning to receive Epo or Darbe during hospitalization
* Infants in whom no aggressive therapy is planned
* Family will NOT be available for follow-up at 22-26 months

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 650 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2025-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Ohls, MD, Principal Investigator — University of Utah
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov) or NHLBI BIOLINCC (https://biolincc.nhlbi.nih.gov/home/).

REFERENCES:
- [Derived] Maxwell JR, Ohls RK, An G, Winter D, Beauman S, Buhrman J, Jantzie LL. Development of an electrochemiluminescence assay to measure serum darbepoetin concentration in extremely preterm infants. Bioanalysis. 2025 Dec 14:1-7. doi: 10.1080/17576180.2025.2600914. Online ahead of print. PMID 41392547
- [Derived] Ohls RK, Das A, Tan S, Lowe JR, Schibler K, Beauman SS, Bell EF, Laptook AR, Baserga M, Patel RM, Carlton DP, Flibotte J, Grisby C, Higgins RD, Shankaran S, Watterberg K, Hibbs AM, Carlo WA, Colaizy TT, Van Meurs KP, Kicklighter SD, Moore R, Sollinger C, Chalak LF, Ghavam S, Poindexter BB, Tyson JE, Cotten CM, Baack ML, Fathi O, DeMauro SB, Laughon MM, Reynolds AM, Duncan AF, Winter S, Wilson-Costello DE, Peralta-Carcelen M, Vohr BR, Harmon HM, Hintz SR, Cavanaugh B, Heyne RJ, Merhar S, Mosquera R, Sewell E, Malcolm WF, Richards LA, Benninger KL, Trembath A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Darbepoetin, Red Cell Mass, and Neuroprotection in Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2025 Aug 1;179(8):836-845. doi: 10.1001/jamapediatrics.2025.0807. PMID 40354084
- [Derived] Bahr TM, Tan S, Smith E, Beauman SS, Schibler KR, Grisby CA, Lowe JR, Bell EF, Laptook AR, Shankaran S, Carlton DP, Rau C, Baserga MC, Flibotte J, Zaterka-Baxter K, Walsh MC, Das A, Christensen RD, Ohls RK; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Serum ferritin values in neonates <29 weeks' gestation are highly variable and do not correlate with reticulocyte hemoglobin content. J Perinatol. 2023 Nov;43(11):1368-1373. doi: 10.1038/s41372-023-01751-z. Epub 2023 Aug 18. PMID 37596391
- [Derived] Vu PT, Ohls RK, Mayock DE, German KR, Comstock BA, Heagerty PJ, Juul SE; PENUT Consortium. Transfusions and neurodevelopmental outcomes in extremely low gestation neonates enrolled in the PENUT Trial: a randomized clinical trial. Pediatr Res. 2021 Jul;90(1):109-116. doi: 10.1038/s41390-020-01273-w. Epub 2021 Jan 11. PMID 33432157

RESULTS

PARTICIPANT FLOW:
Groups:
- Darbepoetin: Darbepoetin (Amgen, Thousand Oaks, CA), 10 mcg per kg, administered once weekly from 36 hours of birth through 35 weeks' PMA, intravenously when the infant had intravenous access, otherwise subcutaneously
- Placebo: Normal saline, 0.4 mL/kg, administered once weekly from 36 hours of birth through 35 weeks' postmenstrual age as a sham subcutaneous dose
Period: Overall Study
Arm/Group | Darbepoetin | Placebo
Started | 322 | 328
Completed Assessment for Bayley Cognitive Score at Two-Year Follow-Up | 239 | 239
Died After Hospital Discharge | 2 | 3
Died Before Hospital Discharge | 50 | 50
Started Study Drug and Data Not Withdrawn Prior to Hospital Discharge | 316 | 325
Survived to Hospital Discharge (a Median of 94 Days) | 269 | 277
Completed (Complete data for Primary Outcome, Bayley Cognitive Score assessed at Two-Year Follow-up, with imputed scores for deaths occurring prior) | 291 | 292
Not Completed | 31 | 36
Not completed — Incomplete Follow-up | 10 | 15
Not completed — Lost to Follow-up | 18 | 20
Not completed — Data withdrawn prior to hospital discharge | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Darbepoetin: Darbepoetin (Amgen, Thousand Oaks, CA), 10 mcg per kg, administered once weekly from 36 hours of birth through 35 weeks PMA, intravenously when the infant had intravenous access, otherwise subcutaneou
- Placebo: Normal saline, 0.4 mL/kg, administered once weekly from 36 hours of birth through 35 weeks postmenstrual age as a sham subcutaneous dose
- Total: Total of all reporting groups
Arm/Group | Darbepoetin | Placebo | Total
Number analyzed (Participants) | 322 | 328 | 650
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age refers to the infant and is measured as gestational age in weeks
  weeks | 26.2 (1.7) | 26.2 (1.6) | 26.2 (1.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 166 | 162 | 328
  Male | 156 | 166 | 322
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 56 | 110
  Not Hispanic or Latino | 263 | 265 | 528
  Unknown or Not Reported | 5 | 7 | 12
Birth weight, Continuous [Mean (Standard Deviation); unit: grams] | 838.2 (252.9) | 822.1 (238.5) | 830.1 (245.7)
Race, Customized [Count of Participants; unit: Participants] — The subject's race is derived from the race of the biological mother
  Participants
    American Indian or Alaska Native | 7 | 11 | 18
    Asian, Native Hawaiian, or Other Pacific Islander | 15 | 7 | 22
    Black or African American | 96 | 102 | 198
    More Than One Race | 7 | 2 | 9
    Unknown or Not Reported | 7 | 9 | 16
    White | 190 | 197 | 387

OUTCOME MEASURES:

1. Primary Outcome: Bayley III Composite Cognitive Score
Description: Bayley Scale of Infant and Toddler Development (BSID)-III composite cognitive score, where subjects who died prior to the follow-up assessment are assigned the lowest possible score of 54. This is a standardized scale where a score that is more than 1 normative standard deviation from the normative mean of 100 signifies mild developmental delay (score < 85); 2 standard deviations below the mean, moderate delay (score < 70); and 3 standard deviations below the mean, severe delay (score < 55). This self-standing scale comprises the primary outcome for the Darbe study.
Time Frame: 22-26 months corrected age (a median of 25 months corrected age, which corresponds to a median of 29 months calendar age in the analysis population), unless the subject died earlier
Population: The analysis population includes all randomized infants with available data up to the two-year followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 291 | 292
score on a scale | 80.7 (19.5) | 80.1 (18.7)
Statistical Analysis 1: Comparison: Darbepoetin vs Placebo; Null hypothesis: Weekly administration of Darbepoetin during the neonatal period will not impact neurocognitive outcomes at 22-26 months compared to Placebo in premature infants 23 to 28 weeks gestation; Test type: Superiority; p = 0.88, Mixed Models Analysis — The mean difference in Bayley-III cognitive scores between treatment groups was adjusted for center, gestational age group, and familial clustering; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-3.09 to 2.64] — Adjusted mean difference in cognitive score for the Darbepoetin minus Placebo treatment groups

2. Secondary Outcome: Number of Transfusions Per Infant
Description: The number of transfusions recorded during the study, up to 35 completed weeks gestational age
Time Frame: Birth, up to the earliest of: death, hospital discharge, or 35 completed weeks gestational age (a median of 9 weeks)
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Mean (Standard Deviation); unit: Transfusions
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 319 | 327
Transfusions | 2.3 (3.1) | 3.3 (3.5)

3. Secondary Outcome: Total Volume of Transfusions Per Infant
Description: The total volume of transfusions for the infant if ever transfused
Time Frame: Birth, up to the earliest of: death, hospital discharge, or 35 completed weeks gestational age (a median of 9 weeks)
Population: The analysis population includes all randomized infants that were ever transfused.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 192 | 257
mL | 54.5 (51.9) | 69.0 (51.0)

4. Secondary Outcome: Number of Donor Exposures Per Infant
Description: The number of donor exposures recorded during the study, up to 35 completed weeks gestational age
Time Frame: Birth, up to the earliest of: death, hospital discharge, or 35 completed weeks gestational age (a median of 9 weeks)
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Mean (Standard Deviation); unit: Donors
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 319 | 327
Donors | 1.6 (2.3) | 2.2 (2.3)

5. Secondary Outcome: Hematocrit
Description: Hematocrit adjusted for center, gestational age group, and familial clustering
Time Frame: at 2 and at 7 weeks in the study
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of blood volume made up of RBCs
Groups:
- Darbepoetin: Darbepoetin (Amgen, Thousand Oaks, CA), 10 mcg per kg, administered once weekly from 36 hours of birth through 35 weeks postmenstrual age, intravenously when the infant had intravenous access, otherwise subcutaneously
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 314 | 319
Percent of blood volume made up of RBCs
  week 2: number analyzed (Participants) | 290 | 292
  week 2 | 36.84 [36.35 to 37.33] | 33.88 [33.4 to 34.36]
  week 7: number analyzed (Participants) | 250 | 266
  week 7 | 37.02 [36.45 to 37.59] | 31.78 [31.24 to 32.32]

6. Secondary Outcome: Red Cell Mass
Description: Red Cell Mass (Circulating Erythrocyte Volume), adjusted for center, gestational age group, and familial clustering
Time Frame: at 2 and at 7 weeks in the study
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 319 | 327
mL
  week 2: number analyzed (Participants) | 305 | 307
  week 2 | 28.35 [27.26 to 29.43] | 24.74 [23.67 to 25.82]
  week 7: number analyzed (Participants) | 272 | 280
  week 7 | 42.78 [41.65 to 43.92] | 36.01 [34.9 to 37.12]

7. Secondary Outcome: Necrotizing Enterocolitis, Bells Stage >=2 With Surgery
Description: This is measured as Yes if experienced necrotizing enterocolitis, Bells stage >=2 with surgery; Otherwise, No.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 94 days)
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 319 | 327
Participants
  Necrotizing Enterocolitis with Surgery | 14 | 13
  No Necrotizing Enterocolitis with Surgery | 305 | 314

8. Secondary Outcome: Bronchopulmonary Dysplasia Grades 2 or 3
Description: This is measured as Yes if infant is on invasive mechanical ventilation, nasal cannula >2 L/min or noninvasive positive airway pressure at 36 weeks of postmenstrual age; Otherwise, No.
Time Frame: At 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 261 | 277
Participants
  Bronchopulmonary Dysplasia at 36 Weeks Postmenstrual Age | 91 | 128
  No Bronchopulmonary Dysplasia at 36 Weeks Postmenstrual Age | 170 | 149

9. Secondary Outcome: Retinopathy of Prematurity Stage >=3 or Treatment for That Condition Received
Description: This is measured as Yes if experienced Retinopathy of prematurity stage >=3 or treatment for that condition received; Otherwise, No. Higher stages of ROP indicate a worse outcome; the stages range from 1 for "mild" disease, to 5 for "severe" disease.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 94 days)
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 273 | 279
Participants
  No Retinopathy of Prematurity Stage At least stage 3 or Treatment for That Condition Received | 238 | 234
  Retinopathy of Prematurity At least stage 3 or Treatment for That Condition Received | 35 | 45

10. Secondary Outcome: Intraventricular Hemorrhage Grade I+
Description: This is measured as Yes if experienced Grade I+ Intraventricular Hemorrhage; Otherwise, No.
Time Frame: Birth to initial hospital discharge or to death if it occurs earlier (a median of 94 days)
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 315 | 318
Participants
  Grade 1+ Intraventricular Hemorrhage | 108 | 98
  No Intraventricular Hemorrhage | 207 | 220

11. Secondary Outcome: Length of Hospital Stay
Description: This is measured as the length of stay up to hospital discharge or death, whichever occurred first.
Time Frame: At initial hospital discharge or at death if it occurs earlier (a median of 94 days), assessed up to one year of life.
Population: The analysis population includes all randomized infants with available data during the initial hospitalization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 304 | 318
Days | 96.2 (58.5) | 104.8 (67.3)

12. Secondary Outcome: Death
Description: This is measured as Yes if an infant died between birth and 22-26 months corrected age; Otherwise, No.
Time Frame: Birth, through the 22-26 months corrected age follow-up window, which corresponds to a median of 29 months calendar age in the analysis population
Population: The analysis population includes all randomized infants with available data up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 319 | 327
Participants
  Death | 52 | 53
  No Death | 267 | 274

13. Secondary Outcome: Neurodevelopmental Impairment
Description: This is a 4-level outcome, where Severe NDI denotes a BSID III cognitive score less than 70, a Gross Motor Functional (GMF) level of 3-5 (where higher scores indicate worse outcomes), blindness (less than 20/200 vision), and/or profound hearing loss, Moderate NDI denotes a BSID III cognitive score from 70-84 and either a GMF level of 2 or limited blindness / moderate hearing loss, Mild NDI denotes a BSID III cognitive score from 70-84, or a cognitive score >=85 with a GMF level of 1 and/or mild hearing loss, and No NDI denotes a cognitive score >= 85 and an absence of neurosensory deficits.
Time Frame: At 22-26 months corrected age (a median of 25 months corrected age)
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 231 | 237
Participants
  Mild | 72 | 68
  Moderate | 1 | 3
  None | 121 | 124
  Severe/profound | 37 | 42

14. Secondary Outcome: Any Cerebral Palsy
Description: This is measured as Yes if the child has been deemed by the medical examiner as having Cerebral Palsy; Otherwise, No.
Time Frame: At 22-26 months corrected age (a median of 25 months corrected age)
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin | Placebo
Number analyzed (Participants) | 244 | 247
Participants
  Any Cerebral Palsy | 40 | 38
  No Cerebral Palsy | 204 | 209

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs were monitored from the first dose of study drug through 36 completed weeks PMA (7 days after administration of the last dose of study drug). All-cause mortality was monitored through 22-26 months corrected age.
Description: Denominators for SAEs and Other AEs were set to the number of randomized subjects who started study drug and did not withdraw from the study prior to hospital discharge. Thus, a total of 9 randomized subjects (5 who never started study drug, and an additional 4 who withdrew from the study prior to discharge) were excluded from these denominators. The denominator for all-cause mortality is the randomized population, excluding the four subjects that withdrew from the study prior to discharge.
Arm/Group | Darbepoetin | Placebo
All-Cause Mortality (participants affected / at risk) | 52/319 | 53/327
Serious Adverse Events (participants affected / at risk) | 85/316 | 92/325
Other Adverse Events (participants affected / at risk) | 16/316 | 21/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin (N=316) | Placebo (N=325)
Acute anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
DIC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Twin-twin transfusion syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Congenital anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 7 (7) | 13 (13)
Neonatal intestinal perforation (Gastrointestinal disorders) | 11 (11) | 12 (12)
Pneumoperitoneum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Direct hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 2 (3)
Failure liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Neonatal sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 32 (34) | 26 (27)
Staphylococcus aureus pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrospinal fluid volume increased (Investigations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular hemorrhage neonatal (Nervous system disorders) | 6 (6) | 4 (4)
Posthaemorrhagic hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 2 (2)
Extreme immaturity (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory decompensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syndrome respiratory distress newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension neonatal (Vascular disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Thrombosis (Vascular disorders) | 4 (4) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin (N=316) | Placebo (N=325)
Sepsis neonatal (Infections and infestations) | 16 (18) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03169881/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03169881/SAP_001.pdf